CLINICAL TRIAL: NCT03178136
Title: HR-HPV Multi-site Opportunistic Screening in Liaoning, China
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Min Wang (Other)
Collaborators: First Hospital of China Medical University (Other); Shenyang women's and children's hostipal (Unknown); Dalian Medical University (Other); The Second Affiliated Hospital of Dalian Medical University (Other); Dandong women's and children's hostipal (Unknown); The First People's Hospital of Jingzhou (Other); The second hospital of Chaoyang City (Unknown); Women's and children's hospital of Yingkou City (Unknown); Cancer hospital of Anshan City (Unknown); Hangzhou Dalton Biosciences,LtD (Unknown)
Responsible Party: Sponsor-Investigator, Min Wang, professor, Shengjing Hospital
Organization: Shengjing Hospital (Other)
Other Study IDs: LSBCIGO-1-DH3-2016-12
Record Dates: First submitted 2017-05-20; First posted 2017-06-06 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2019-01

CONDITIONS: Cervical Cancer
Keywords: HR-HPV opportunistic screening; virus load; multi-site
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — cervical cell
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- case group: There is no intervention in case group.
- control group: The control group as the contrast for case group.

SUMMARY:
It is universally accepted that the persistent infection of high-risk human papillomavirus(HR-HPV) is the cause of cervical intraepithelial neoplasias and cancer. Some researches indicate that the virus load may relate the extent of the disease. The objective of the study is to detect the virus load of 14 types HR-HPV among the participants, using a new HPV DNA hybrid capture technology,sequentially find the diagnostic significance of virus load of HPV.

DETAILED DESCRIPTION:
Cervical cancer is the most common malignancy in women, the persistent infection of high-risk human papillomavirus(HR-HPV) is the definite cause,especially the infection of human papillomavirus 16/human papillomavirus 18(HPV16/HPV18). Some researches indicate the virus load may relate the extent of the disease, but the sample capacity is not enough to receive a conclusive conclusion. And a specific quantity or a range of virus load which closely relates to cervical intraepithelial neoplasia 2(CIN2) or worse is not studied. The aim of the study is to prove the association between the virus load and development of cervical intraepithelial neoplasias by detecting 14 types HR-HPV, and find the specific quantitative value or the range to assist physician to diagnose.

A detect reagent named Dalton hybrid 3(DH3) is used in the study, the mechanism of which is HPV DNA hybrid capture technology, the experimental process include seven steps, denaturation, hybridization, the formation of DNA-RNA heterozygote, capture, detect, rinse panel, read data.

Study design: The organizations of the study contain ten hospitals in Liaoning province in China,patients accord with inclusion criteria(N=10000) sign informed consent and fill out a information form. Gynecologist collect cervical cell with sampling instrument. Detecting the virus load of HPV16/HPV18 and other 12 types HR-HPV, the positive result is cut-off ≥1.0pg/ml, HPV16/HPV18(+) need colposcopy. The abnormal result of colposcopy requires biopsy, the participant who has abnormal result of biopsy need operative treatment. Follow-up observation of all participants lasting 5 years are required.

ELIGIBILITY:
Inclusion Criteria:

The patients who are voluntary to accept screening with sexual life

Exclusion Criteria:

uterectomy, cancer, other serious illness, physical examination(pregnant women are not exclusive)

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients who are voluntary to accept screening with sexual life between the age of 25 to 65 are the target population of the study.
  The population who with uterectomy, cancer, other serious illness, physical examination are exclusive, the pregnant women are not exclusive.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2017-06-19 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
virus load | 1 day
  virus load of 14 types HR-HPV

CONTACTS AND LOCATIONS:
Overall Officials: Min Wang, Study Director — Shengjing Hospital
Locations (7):
- China (7):
  - Cancer hospital of Anshan City, Anshan, Liaoning
  - The second hospital of Chaoyang City, Chaoyang, Liaoning
  - Dalian obstetrics and gynaecology hospital, Dalian, Liaoning
  - The first affiliated hospital of Jinzhou Medical University, Jinzhou, Liaoning
  - The first hospital of China Medical University, Shenyang, Liaoning
  - Women's and children's hospital of Yingkou City, Yingkou, Liaoning
  - Shenyang women's and children's hospital, Shenyang, Lioaning

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Snijders PJ, van den Brule AJ, Meijer CJ. The clinical relevance of human papillomavirus testing: relationship between analytical and clinical sensitivity. J Pathol. 2003 Sep;201(1):1-6. doi: 10.1002/path.1433. PMID 12950011
- [Background] Vorsters A, Van Keer S, Biesmans S, Hens A, De Coster I, Goossens H, Ieven M, Van Damme P. Long-Term Follow-up of HPV Infection Using Urine and Cervical Quantitative HPV DNA Testing. Int J Mol Sci. 2016 May 17;17(5):750. doi: 10.3390/ijms17050750. PMID 27196899
- [Result] Wakeham K, Kavanagh K, Cuschieri K, Millan D, Pollock KG, Bell S, Burton K, Reed NS, Graham SV. HPV status and favourable outcome in vulvar squamous cancer. Int J Cancer. 2017 Mar 1;140(5):1134-1146. doi: 10.1002/ijc.30523. PMID 27864932
- [Derived] Wang M, Hou B, Wang X, Han L, Shi Y, Zhang Y, Zhang L, Liu L, Jin F, Zhang Y. Diagnostic value of high-risk human papillomavirus viral load on cervical lesion assessment and ASCUS triage. Cancer Med. 2021 Apr;10(7):2482-2488. doi: 10.1002/cam4.3653. Epub 2021 Mar 7. PMID 33682355